CLINICAL TRIAL: NCT01073982
Title: Efficacy of Tart Cherry Juice to Reduce Pain and Inflammation Among Patients With Inflammatory Osteoarthritis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: Cherry Research Committee (Other)
Responsible Party: Kerry S. Kuehl MD PhD/Associate Professor, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: e5825
Record Dates: First submitted 2010-02-12; First posted 2010-02-24 (Estimated); Last update posted 2011-01-20 (Estimated); Status verified 2011-01

CONDITIONS: Pain; Inflammation
Keywords: pain; inflammation; osteoarthritis
MeSH Terms: conditions — Pain; Inflammation; Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- cherry flavored fruit drink (Placebo Comparator)
  Interventions: Dietary Supplement: tart cultivar Montmorency cherry juice
- tart cherry juice (Experimental)
  Interventions: Dietary Supplement: tart cultivar Montmorency cherry juice

INTERVENTIONS:
Dietary Supplement: tart cultivar Montmorency cherry juice — 21 ounces of experimental or placebo juice, consumed daily for 21 days.

SUMMARY:
The purpose of this study is to assess the effects of tart cherry juice to reduce pain and inflammation among individuals with arthritis.

DETAILED DESCRIPTION:
Numerous antioxidant and anti-inflammatory agents have been identified in tart cherries, and a study among healthy, non-exercising individuals demonstrated that cherry consumption decreased serum inflammatory biomarkers after 14 days. Osteoarthritis (OA) is a common syndrome affecting 65 million Americans characterized by pain, inflammation, and disability. Such natural anti-inflammatory effects of cherry consumption may be beneficial for the management and treatment of osteoarthritis and inflammatory diseases. The purpose of this randomized, double-blind, placebo controlled study is to examine individuals with inflammatory OA and assess the analgesic and anti-inflammatory effects of tart cherry juice as compared to a placebo drink among twenty 30-70 y/o OA subjects.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with inflammatory osteoarthritis
* In good general health
* Stable pattern of anti-inflammatory or pain relieving drug use for 3 months prior to study
* Ability and willingness to maintain consistent pattern of anti-inflammatory or pain relieving drug use during the course of the study, and to not seek any other treatment during the study
* Ability and willingness to consume juice or placebo drink for 21 consecutive days, and to participate in screening measures, including a blood draw, before and after the intervention period

Exclusion Criteria:

* Pregnancy
* Serious medical conditions such as recent heart attack or stroke, cancer, diabetes (type 1 and type 2), or gastrointestinal ulcers
* Individuals who have not been on a stable dose of pain medications or pain modalities for at least 3 months, including muscle relaxants, tender point anesthetic injections, systemic or intrabursal or intraarticular steroids, or any investigational drug/device in the prior 90 days
* Individuals who have used nonpharmacologic pain therapies including acupuncture, ultrasound, or transcutaneous electrical nerve stimulation within the past 30 days

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2010-02; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Primary outcomes include measurement of interleukin 10 (IL-10), CRP, and a specific group of cytokines that provide a generalized measurement of inflammatory activity, these include IL-6 and TNF-α. | 6-8 months

CONTACTS AND LOCATIONS:
Overall Officials: Kerry S Kuehl, MD, PhD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health and Science University, Portland, Oregon, United States